CLINICAL TRIAL: NCT03088735
Title: Pilot Study of the Best Transfer Strategy in an Oocyte Donation Programme: an Intention to Treat Randomized Controlled Trial
Brief Title: Transfer Strategy in an Oocyte Donation Programme
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the clinically and statistically significant inferior results for the D3 group following evaluation by the institutional review board.
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Elisabet Clua Obrado, Head of Gamete and Embryo Donation, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMD-2017-03
Record Dates: First submitted 2017-03-18; First posted 2017-03-23 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Oocyte Donation; Infertility, Female; Embryo Transfer
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blastocyst-stage embryo transfer strategy (Experimental)
  Interventions: Procedure: Blastocyst-stage embryo transfer strategy
- Cleavage-stage embryo transfer strategy (Active Comparator)
  Interventions: Procedure: Cleavage-stage embryo transfer strategy

INTERVENTIONS:
Procedure: Blastocyst-stage embryo transfer strategy — Intra-uterine transfer of blastocist if in cleavage embryo stage the oocyte recipient has a mínimum of 3 availables embryos with at least one of good quality to transfer and also the inta-uterine transfer of cleavage embryo (day 3) when the recipient doesn't have the previous criteria.
  Arms: Blastocyst-stage embryo transfer strategy
Procedure: Cleavage-stage embryo transfer strategy — Inta-uterine transferring of cleavage embryo transfer (day 3 of develpment) in oocyte recipients
  Arms: Cleavage-stage embryo transfer strategy

SUMMARY:
It has been previously shown that although the activation of the embryonic genome can begin as early as two days of initiation of the embryonic development (D2), it is expressed on day 3 (D3). Without this activation, the embryo can not continue its development. Therefore, it has been suggested that extended culture to blastocyst stage could be an option to identify and better select embryos that have been able to carry out this activation. The purpose of this study is to compare cumulative pregnancy and live birth rates following transfer of cleavage embryos or blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* Patients under their first or second cycle of a synchronous (fresh) oocyte donation cycle.

Exclusion Criteria:

* Preimplantation genetic screening or diagnosis cycles.
* Patients with strict blastocyst-stage embryo transfer indication by the couple's treating physician.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 134 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Cumulative live birth rate | at 12 months after a embryo transfer (time considered enough in order to do a minimum of one frozen-thawed cycle if pregnancy is not achieved with the fresh cycle
  Total number of births considering fresh and frozen thawed embryos transferred

SECONDARY OUTCOMES:
Cumulative pregnancy rate | at 12 months after a embryo transfer (time considered enough in order to do a minimum of one frozen-thawed cycle if pregnancy is not achieved with the fresh cycle
  Total number of pregnancies confirmed by ultrasound 6 weeks after embryo transfer including fresh and thawed embryos.

CONTACTS AND LOCATIONS:
Locations (1):
- Department Obstetric, Gynecologic and Reproductive Medicine, Barcelona, Barcelons, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.dexeus.com